CLINICAL TRIAL: NCT04452604
Title: National Retrospective Monitoring of Patients With Acute Leukemia Infected by COronaVirus Disease 2019 (COVID-19)
Brief Title: Multicentric Registry of Patients With Acute Leukemia Infected by COVID-19
Acronym: COVLA
Status: Completed | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Acute Leukemia French Association (Other); Group for Research in Adult Acute Lymphoblastic Leukemia (Other)
Responsible Party: Sponsor
Other Study IDs: COVLA
Record Dates: First submitted 2020-06-18; First posted 2020-06-30 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Acute Myeloblastic Leukemia; Acute Lymphoblastic Leukemia; SARS-CoV-2
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 epidemic (Coronavirus Disease 2019) currently raging in France is an emerging infectious disease linked to a virus of the genus coronavirus (SARS-CoV-2). Epidemiologically, acute myeloblastic leukemias (AML) are the most common of acute leukemias. The incidence of acute lymphoblastic leukemia (ALL) is 900 new cases in France in 2018, of which 57% in humans. The treatments administered to AML and ALL patients induce variable immunosuppression: neutropenia, neuropathy, deficits in humoral or cellular immunity or combinations of these deficits. Patients with AML or ALL therefore represent a population at high risk of developing a serious form in the event of infection with SARS-CoV-2. To date, no data is available in the literature to assess the impact of the COVID-19 epidemic in the population of patients with acute leukemia.

The main objective of the study is to determine the clinical and biological prognostic factors during SARS-CoV-2 infection in patients with acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute leukemia according to WHO criteria 2016 ≤ 5 years
* Diagnosis of a proven or probable SARS-CoV-2 infection according to the following criteria:

  1. Proven infection: positive Polymerase Chain Reaction (PCR) regardless of the radio-clinical picture (other tests made available later and having good diagnostic performance will be accepted)
  2. Probable infection: negative PCR but association of

     1. Evocative clinical signs, of recent installation: fever, respiratory signs (cough, dyspnea, chest pain), body aches, sore throat, rhinorrhea, headache, diarrhea / abdominal pain, frank asthenia, loss of taste / smell, conjunctivitis, type of frostbite AND
     2. evocative radiological signs, on CT: diffuse or diffuse aspect of frosted glass, condensations including pseudo-nodular condensations, association of frosted glass and condensation within the same lesion, nodules and micronodules, thickening of the interlobular septa) or on chest radiography: interstitial, alveolo-interstitial or alveolar syndrome, single or bilateral AND
     3. absence of differential diagnosis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 infected patients with AML or ALL
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Clinical prognostic factors for infection with COVID-19 | Day 0
  Factors associated with overall survival will be analyzed : center, sex, leukemia subtype, previous treatment by corticosteroids, and comorbidities (respiratory, renal, cardiac, weight, diabetes)
Biological prognostic factors for infection with COVID-19 | Day 0
  neutrophils and lymphocytes count at the time of SARS-COV2 infection
Medical care of Coronavirus infection | within 12 months after diagnosis
  Describe the management carried out concerning coronavirus infection and its impact of the treatment of acute leukemia (non-invasive ventilation, orotracheal intubation, vasopressor requiring, treatments used, cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves DUMAS, Dr, Principal Investigator — French Innovative Leukemia Organisation
Locations (27):
- France (27):
  - Chu Amiens, Amiens
  - CHU ANGERS - Maladies du sang, Angers
  - Ch Avignon, Avignon
  - CH de la Côte Basque - Hématologie, Bayonne
  - CHU Caen - IHBN - Hématologie Clinique, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier de Dunkerque, Dunkirk
  - CHU de Grenoble - Hopital Michallon, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital Saint Vicent de Paul, Lille
  - Chu Limoges, Limoges
  - Institut Paoli-Calmettes - Hématologie 2, Marseille
  - HOPITAL SAINT ELOI - Hematologie, Montpellier
  - HOPITAL E. MULLER - Hématologie, Mulhouse
  - CHU HOTEL DIEU - Hématologie Clinique, Nantes
  - CHU Caremeau, Nîmes
  - CENTRE HOSPITALIER SAINTJEAN - Hématologie Clinique, Perpignan
  - Bordeaux Pessac, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Reims - Hôpital Robert Debré - Hématologie Clinique, Reims
  - CHU Pontchaillou - Hématologie, Rennes
  - Chu de La Reunion - Site Sud, Saint-Pierre
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Universitaire du Cancer de Toulouse Oncopole - Service d'Hématologie, Toulouse
  - CHU de Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier de Versailles, Versailles
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No